CLINICAL TRIAL: NCT01799759
Title: Project Fun: Parents And Youth Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HR-1625
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Childhood Obesity
Keywords: Body Mass Percentile; Authoritative parenting; Online interventions; Prevention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online intervention for parent and child (Experimental): Children complete 8 online modules of Project FUN Parents complete 6 modules of Project FUN for Parents
  Interventions: Behavioral: Online intervention
- Instruments only (Other): The waiting list control group only completes instruments and body composition, fitness measures
  Interventions: Other: Completion of instruments only

INTERVENTIONS:
Behavioral: Online intervention — Child online intervention is 8 modules based on the Health Promotion/Transtheoretical Model Parent online intervention is 6 modules based on enhancing authoritative parenting,support and role models for improved nutrition, physical activity and health child body mass percentile
  Arms: Online intervention for parent and child
Other: Completion of instruments only — Parent and child subejects in the waiting list control only complete surveys, body composition and fitness tests
  Arms: Instruments only

SUMMARY:
The proposed study is a continuation of a randomized, controlled pilot effectiveness trial conducted in schools wherein the feasibility and completion of the trial by parents and children will now additionally be examined in after school and YMCA connected programs.

The intervention for this study is Project FUN and Project FUN with Parents. Project FUN is an 8 module online program for children in 4th through 8th grade. Project FUN with Parents is a 6 module online program for their parent.

Children and parents will be recruited through the afterschool and YMCA connected programs. Those agreeing to participate will be randomly assigned to a first intervention or second intervention session (waiting list control group). Surveys and measures will be collected for everyone pre-intervention, after the first session completion and after the second session completion to create a waiting list control group.

Hypothesis 1: Body composition and dietary fat of children who complete Project FUN and have a parent complete Project FUN with Parents will be lower on completion than children who only complete instruments.

Hypothesis 2: Fruit and vegetable intake, physical activity and fitness of children who complete Project FUN and have a parent complete Project FUN with Parents will be greater on completion than children who only complete instruments.

DETAILED DESCRIPTION:
Addressing the epidemic of obesity is a national priority. Currently almost a third of children and two thirds of adults are overweight or obese. Obesity-related chronic health problems originating in childhood are often life-long. Overweight and obesity result from detrimental patterns of dietary intake and physical activity. These obesity-producing lifestyles are established in childhood and are often carried into adulthood, when they become more refractory to change. Research has demonstrated that programs involving parents and children in a family context have been the most effective in preventing and treating childhood obesity.

Research Question 1: How many parents and children agree to participate, complete data collection and complete at least 80% of the intervention? Research Question 2: What reasons are given by those not completing the protocol and what suggestions are offered by those who do complete the protocol? Research Question 3: What is the relationship of parent or child perceptions of authoritative parenting, child perceptions of family models and support for healthy eating, physical activity, or reduced sedentary time, and of parenting stress, self-efficacy, confidence, and eating behavior on child BMI? Research Question 4: Do parent or child perceptions of authoritative parenting, diet, physical activity, fitness or body composition; child perceptions of family models and support for healthy eating, physical activity, or reduced sedentary time; or parent perceptions of parenting stress, self-efficacy, confidence, and eating behavior change across the study time period? Research Question 5: Are there relationships between study completion and child or parent BMI, child or parent gender, parenting stress, self-efficacy, confidence, and eating behavior?

ELIGIBILITY:
Inclusion Criteria:

* Children in 4th through 8th grade and a parent(s)who can read and write English. Must be able to come to Marquette University or Milwaukee area YMCA for pre and post test data collection and to complete online modules.

Exclusion Criteria:

* None

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
child body mass percentile | 6-12 weeks
  Child height and weight are measured and the body mass percentile calculated using the Centers for Disease Control and Prevention algorithm for adjustment by age and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Frenn, PhD, RN, Principal Investigator — Marquette University College of Nursing
Locations (1):
- Marquette University College of Nursing, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No